CLINICAL TRIAL: NCT00217139
Title: A Phase II, Randomized, Active-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Celgosivir in Combination With Peginterferon Alfa-2b, With and Without Ribavirin, for 12 Weeks in Patients With Chronic Hepatitis C Infection (Genotype 1) Who Failed to Respond to Pegylated α Interferon-Based Therapy
Brief Title: A Study to Evaluate the Safety and Efficacy of Celgosivir and Peginterferon Alfa-2b, With or Without Ribavirin, in Patients With Chronic Hepatitis C Genotype 1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioWest Therapeutics Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV-05-002
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-09-29 (Estimated); Status verified 2006-09

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; Celgosivir; HCV; Genotype 1; Non-responders; Early Viral Response; EVR
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — celgosivir

INTERVENTIONS:
Drug: Celgosivir

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of celgosivir plus peginterferon alfa-2b, with or without ribavirin, for 12 weeks in patients with chronic hepatitis C genotype 1 infection.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, inclusive
* primary diagnosis of chronic HCV infection
* non-responders to previous pegylated interferon-based therapy

Exclusion Criteria:

* patients naive to interferon-based therapy for chronic HCV infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-09; Study Completion 2006-09

PRIMARY OUTCOMES:
Safety analysis
HCV viral load

CONTACTS AND LOCATIONS:
Overall Officials: Jim Pankovich, Study Director — BioWest Therapeutics Inc
Locations (6):
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario